CLINICAL TRIAL: NCT05506462
Title: An Open Label Study of Electroencephalographic Responses Pre, During and Post, a Low Dose, Weekly Intravenous Ketamine Infusion for 4 Weeks, in a Study Population With Major Depression Disorder
Brief Title: An EEG Study of Intravenous Ketamine for Major Depression Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ehave Inc. (Industry)
Collaborators: Tristar Wellness (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21EERPZ01
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder
Keywords: Intravenous ketamine; Electroencephalogram (EEG) monitoring; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine (Experimental): 50-60 minutes intravenous infusion of 60mg ketamine
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Patients with a diagnosis of Major Depressive Disorder (MDD) will be enrolled to receive four 50-60 minute infusions of 60mg ketamine hydrochloride
  Other Names: NDC 67457-108-00

SUMMARY:
There are many common pharmacological treatments for major depression disorder (MDD), however the efficacy of these drugs often fails in severe cases. Intravenous (IV) administered ketamine may offer the potential for remission of the symptoms in patients with MDD; however it has not yet been approved by FDA for this purpose. This study will make use of an electroencephalography (EEG) machine to measure the brain's activity and response while the IV ketamine is being delivered. The objective of this study is to characterize the change in EEG response of patients with MDD, during and 4 weeks after a course of IV ketamine infusions.

DETAILED DESCRIPTION:
This study will enroll 35 patients with major depressive disorder. Candidates for participation in the study will typically be either referred to the clinic through their healthcare provider or will have sought out participation on their own accord based on advertising. Subjects will be screened for eligibility and suitable patients will be invited to attend a screening visit in the clinic and complete informed consent.

Upon determining eligibility, subjects will have their first treatment session booked within 42 days of screening (Baseline, visit 0). Three subsequent weekly (±3 days) ketamine therapy treatment sessions will occur on days 7, 14 and 21, for a total of four ketamine infusions over four weeks. All patients will return for a follow-up visit at 4-weeks post final treatment visit, day 49.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between 18 and 70 years of age, inclusive
2. Adult patients with a documented primary Axis I clinical diagnosis meeting criteria from the DSM-V for a major depressive disorder
3. Score of <15 on the DES
4. Moderate to severe symptoms objectively documented using MADRS total score of ≥ 20
5. Ability to maintain scheduled appointments for screenings, 4 treatment visits and follow-up EEG visit.
6. History of major depressive disorder.
7. Females of child-bearing potential who are sexually active must agree to use two forms of contraception. A pregnancy test will be performed before the first treatment.
8. Must have stable residence address, internet and mobile phone.
9. Must speak fluent English.

Exclusion Criteria:

1. Known allergy to ketamine or any other drug used in the study.
2. Use of ketamine in a therapeutic model within the preceding 12 months of the study.
3. Current or any history of schizoaffective disorder(s).
4. Score of ≥ 15 on DES
5. History of illicit active substance abuse or dependence including ketamine as determined on by the SCID-5-CT and/or drug urine screening during study visits.
6. Pregnancy, breastfeeding or desire to become pregnant during the course of the study.
7. Serious, unstable illnesses including, but not limited to; hepatic, gastro-intestinal, respiratory, cardiovascular (including ischemic heart disease and coronary heart disease). History of ischemic stroke, atrial fibrillation, severe endocrinological, neurological, immunological or hematological disease.
8. Any history of cerebral vascular events including stroke, bleeding into the brain and subdural hematomas.
9. Any implantable metallic device(s) or implant(s) above the level of shoulders.
10. Any non-removable metallic piercings.
11. Patients with cochlear implants and non-removable hearing aids.
12. Current use of: Dilantin, Depakote, Phenobarbital, Gabapentin, Pregabalin and Benzodiazepines. Certain candidates with long use of Benzodiazepines may qualify at PI's discretion.
13. Severe labile hypertension.
14. Significant uncontrolled hypertension (i.e., SBP > 150 mmHG, DBP > 100 mmHG)
15. Uncontrolled diabetes mellitus.
16. Patients on renal dialysis.
17. Inability to achieve consistent IV access.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Characterizing the changes in EEG reading frequencies from pre- IV ketamine infusion treatment (baseline). | 30-minute pre-treatment baseline and throughout infusion (approximately 50-60 minutes)
  Alpha, Beta, Delta, Theta and Gamma frequencies will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution
Characterizing the changes in EEG reading waveforms from pre- IV ketamine infusion treatment (baseline). | 30-minute pre-treatment baseline and throughout infusion (approximately 50-60 minutes)
  Alpha, Beta, Delta, Theta and Gamma waveforms will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution
Characterizing the changes in EEG reading amplitudes from pre- IV ketamine infusion treatment (baseline). | 30-minute pre-treatment baseline and throughout infusion (approximately 50-60 minutes)
  Alpha, Beta, Delta, Theta and Gamma amplitude will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution
Characterizing the changes in EEG reading patterns from pre- IV ketamine infusion treatment (baseline). | 30-minute pre-treatment baseline and throughout infusion (approximately 50-60 minutes)
  Alpha, Beta, Delta, Theta and Gamma reading patterns will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution
Characterizing the changes in EEG reading frequencies from pre- IV ketamine infusion treatment (baseline) and 4 weeks post-treatment course | Pre-treatment baseline, 4 weeks post-treatment course
  Alpha, Beta, Delta, Theta and Gamma frequencies will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution
Characterizing the changes in EEG reading waveforms from pre- IV ketamine infusion treatment (baseline) and 4 weeks post-treatment course | Pre-treatment baseline, 4 weeks post-treatment course
  Alpha, Beta, Delta, Theta and Gamma waveforms will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution
Characterizing the changes in EEG reading amplitudes from pre- IV ketamine infusion treatment (baseline) and 4 weeks post-treatment course | Pre-treatment baseline, 4 weeks post-treatment course
  Alpha, Beta, Delta, Theta and Gamma amplitude will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution
Characterizing the changes in EEG reading patterns from pre- IV ketamine infusion treatment (baseline) and 4 weeks post-treatment course | Pre-treatment baseline, 4 weeks post-treatment course
  Alpha, Beta, Delta, Theta and Gamma amplitude will be examined with portable NeuroEEG™, a 19 channels and 22 electrodes cap based on 10-20 distribution

SECONDARY OUTCOMES:
Incidence of medically significant changes in blood pressure during ketamine infusion | Pre-treatment baseline; treatment initiation, 0 minutes; 20 minutes, 40 minutes; 60 minutes post-infusion
Incidence of medically significant changes in Oxygen Saturation (SpO2) during ketamine infusion | Pre-treatment baseline; treatment initiation, 0 minutes; 20 minutes, 40 minutes; 60 minutes post-infusion
Incidence of medically significant changes in heart rate during ketamine infusion | Pre-treatment baseline; treatment initiation, 0 minutes; 20 minutes, 40 minutes; 60 minutes post-infusion
Incidence of medically significant changes in respiratory rate during ketamine infusion | Pre-treatment baseline; treatment initiation, 0 minutes; 20 minutes, 40 minutes; 60 minutes post-infusion
Changes from baseline in the Dissociative Experiences Scale (DES) Total Score | Baseline (Day 0), follow-up visit (Day 42)
  The Dissociative Experiences Scale (DES) is a 28-item scale assessing the subject's experiences in his/her daily life. The subject determines to what degree he/she has been facing the situation by selecting a percentage from 0% (never) to 100% (always), with 10% increments in between. Higher scores mean higher severity

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Kamlet, MD, Principal Investigator — Tristar Wellness

IPD SHARING:
Plan to Share IPD: No